CLINICAL TRIAL: NCT01150331
Title: Efficiency of Levetiracetam Intravenous in Association With Clonazepam Versus Clonazepam Alone in Prehospital Care of Generalised Tonicoclonic Status Epilepticus
Brief Title: Study of Antiepileptic Drug in Generalised Convulsive Status Epilepticus
Acronym: SAMU-KEPPRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P070704
Record Dates: First submitted 2010-04-23; First posted 2010-06-24 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Status; Epilepticus, Tonic-clonic
Keywords: status epilepticus; generalised convulsive status epilepticus; first line treatments; double-blind randomized controlled trial; prehospital treatment
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam; Clonazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonazepam + levetiracetam (Experimental): Clonazepam IV 1 mg+ levetiracetam IV 2500 mg
  Interventions: Drug: Levetiracetam/Clonazepam
- Clonazepam + placebo (Active Comparator): Clonazepam IV 1 mg + placebo levetiracetam IV
  Interventions: Drug: Clonazepam/Placebo levetiracetam IV

INTERVENTIONS:
Drug: Levetiracetam/Clonazepam — Association of two anti-epileptic drugs in first line
  Other Names: Association of two anti-epileptic drugs in first line
  Arms: Clonazepam + levetiracetam
Drug: Clonazepam/Placebo levetiracetam IV — Association of placebo to an active comparator (clonazepam)
  Other Names: Association of placebo to an active comparator (clonazepam)
  Arms: Clonazepam + placebo

SUMMARY:
Compare the efficiency of the association, first line, the intravenous levetiracetam and the intravenous clonazepam, in that of a monotherapy of clonazepam intravenous in the pre-hospital treatment of tonicoclonic generalised status epilepticus.

DETAILED DESCRIPTION:
At this time, the prehospital treatment of the status epilepticus use some molecule ("FOSPHENYLOINE") with large contra-indications. In this case the physician is not able to know the past medical history of the patient, the biological examinations and so he can not decide which molecules he can use.

The levetiracetam is a knowledge medication in the epilepsy since more than twenty years. One of specificity of the levetiracetam is to be able to be used in all situations (no clinical or biological contre-indication). This molecule seems like to be very interesting to be used in prehospital system.

The goal of this study is to evaluate the association levetiracetam / clonazepam in first line in the prehospital treatment of the status epilepticus

ELIGIBILITY:
Inclusion criteria :

* Age ≥ 18 years
* Patient taken care by a prehospital medical team participating in the study
* Diagnosis of tonicoclonic generalized status epilepticus confirmed on the spot by a physician of the team.

Exclusion criteria :

* Parent or the reliable person indicated by the patient present not giving its agreement for the inclusion
* Pregnancy clinically detectable or known for close relations at the time of the status epilepticus
* tonicoclonic generalized status epilepticus after anoxia post cardiac arrest
* Patient having already received another treatment for the same episode of status epilepticus
* Patient having already participated in the study during a previous episode of status epilepticus
* Patient in "latent" status epilepticus. Definition : patient in the coma having epileptic demonstrations (CLONISMS MYOCLONISMS) small or invalid, contrasting with permanent generalized electric seizures on the EEG
* Patient presenting certain diagnosis of pseudo name psychogenic seizure
* Patient whose neurological status requires an immediate surgery (traumatism)
* Patient having a hyper-responsiveness about the levetiracetam or about the other by-products of pyrrolidone or an one of the excipients
* Patient having a hyper-responsiveness about the clonazepam, about the benzodiazepins or about one of the other constituents of the product
* Patient under medical guardianship
* Not membership in a schema of medical assurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-07; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Patient's percentage having stopped convulsing in the 15 minutes following the injection. The stop of the crisis is defined as the stop of all epileptic movements (myoclonic, clonic or tonic) | 15 minutes

SECONDARY OUTCOMES:
Period between the first injection and the clinical stop of the convulsion | up to 15 minutes
Period between the first injection and the presence of signs of awakening | up to three days
Time of hospitalization | up to 15 days
Patient's percentage having received the second injection of clonazepam to T5 min | 5 minutes
Patient's percentage having received an injection of second anticonvulsivant to T15 min | 15 minutes
Patient's percentage presenting signs of awakening to T35 min | 35 minutes
Patient's percentage having been intubated for the general anesthesia | 35 minutes
Score of glasgow coma scale for the patients with no signs of awakening to T35 and to the arrival of the hospital | up to 35 minutes
Patient's percentage having had a recurrence of epileptic seizure during the hospital follow-up | up to 15 days
Patient's percentage presenting convulsions or signs of awakening to the arrival to the hospital | up to 15 days
Frequency of adverse events and their severity | up to 15 days
Frequency of respiratory, hemodynamic and cardiac occurence of complications | up to 15 days
Analysis of the main criteria of efficiency by sous groups according to the etiology of the generalised tonic-clonic status epilepticus and according to this duration during the therapeutic clinical care | up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Carli, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Result] Navarro V, Dagron C, Elie C, Lamhaut L, Demeret S, Urien S, An K, Bolgert F, Treluyer JM, Baulac M, Carli P; SAMUKeppra investigators. Prehospital treatment with levetiracetam plus clonazepam or placebo plus clonazepam in status epilepticus (SAMUKeppra): a randomised, double-blind, phase 3 trial. Lancet Neurol. 2016 Jan;15(1):47-55. doi: 10.1016/S1474-4422(15)00296-3. Epub 2015 Nov 28. PMID 26627366
- [Derived] Navarro V, Dagron C, Demeret S, An K, Lamhaut L, Bolgert F, Baulac M, Carli P. A prehospital randomized trial in convulsive status epilepticus. Epilepsia. 2011 Oct;52 Suppl 8:48-9. doi: 10.1111/j.1528-1167.2011.03236.x. PMID 21967362